CLINICAL TRIAL: NCT00906607
Title: Prevalence of the Urinary Incontinence in Adolescents, Young, Adults and Aged
Brief Title: Prevalence of Urinary Incontinence in Different Age Categories
Status: Completed | Type: Observational
Sponsor: Universidade de Franca (Other)
Responsible Party: Lislei Jorge Patrizzi, Universidade de Franca
Other Study IDs: 0077/08
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group I: 10-18 years
- Group II: 20-35 years
- Group III: 45-60 years
- Group IV: 65-75 years

SUMMARY:
Introduction: Urinary incontinence (UI) is considered erroneously by many as being a phenomenon of the aging process, however there is a growing prevalence of complaints of UI in nulliparous and nulligest young women.

Objective: To investigate the prevalence of urinary incontinence in women of different age groups.

Method: 78 nulliparous and nulligest women of different resident age groups in the city of France, being these divided in: G1 (10-18 years); G2 (20-35 years); G3 (45-60 years) and G4 (65-75 years). Excluded from this study were women with cancer or surgeries of the inferior urinary treatment, urinary infection, alterations cognitive, pregnant and obesity. All the participants were questioned as a perception of urine loss, to the efforts or effortlessly evident.

DETAILED DESCRIPTION:
All participants were asked about perceived loss of urine, the effort or without apparent effort. The responses of participants from G1 were offered by parents and / or responsible.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous and nulligest women

Exclusion Criteria:

* women with cancer reported
* surgeries of the inferior urinary treatment
* urinary infection
* cognitive alterations
* pregnant
* obesity

Ages: 10 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included 78 nulliparous and nulligest women of different ages living in the city of Franca, and these are divided into: G1 (10-18 years), G2 (20-35 years), G3 (45-60 years) and G4 (65-75 years).
  Women with a history of cancer or surgery of the lower urinary tract, urinary tract infection, cognitive changes, pregnancy and obesity, were excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lislei Patrizzi, Study Director — Universidade de Franca